CLINICAL TRIAL: NCT05766111
Title: Seroprevalence Survey in Healthcare Workers of the A. Gemelli IRCCS University Hospital Foundation as Part of the Surveillance and Control Activities of the Covid-19 Epidemic
Brief Title: COVID-19 Seroprevalence Among Healthcare Workers of a Large COVID-19 Hospital in Rome
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Laurenti Patrizia, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3253
Record Dates: First submitted 2023-03-10; First posted 2023-03-13 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Healthcare workers are at the forefront against COVID-19, worldwide. Since Fondazione Policlinico Universitario A. Gemelli (FPG) IRCCS was enlisted as a COVID-19 hospital, the healthcare workers deployed to COVID-19 wards were separated from those with limited/no exposure, whereas the administrative staff were designated to work from home. Between June and July 2020, an investigation will conduct to evaluate the seroprevalence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) immunoglobulin (IgG) antibodies among the employees of the FPG using point-of-care (POC) and venous blood tests. Sensitivity, specificity, and predictive values were determined with reverse-transcription polymerase chain reaction on nasal/oropharyngeal swabs as the diagnostic gold standard.

DETAILED DESCRIPTION:
This cross-sectional study will consist of a seroprevalence survey between June 2020 and July 2020, which enroll participants on a voluntary basis via a hospital e-mail system, including medical, non-medical HCW, and administrative staff (AS) of the FPG. The study approved by the FPG ethics committee and participants sign an informed consent form before their inclusion in the study. Both the venous blood and POC SARS-CoV-2 serological tests will offer to each participant and perform in dedicated blood-drawing areas in compliance with COVID-19 safety regulations. In cases with a positive result from at least one test, participants undergo NOS sampling for RT-PCR SARS-CoV-2 RNA detection to assess the actual infection status . Unlike the venous blood testing, the POC testing will perform by trained clinical staff composed of public health residents and student nurses.Medical and non-medical HCWs will categorize into two groups by whether they had or had not assisted COVID-19 patients in the period between 9 March 2020 (the date of the first COVID-19 patients in our hospital) and 1 June 2020 (the date of seroprevalence survey initiation). For predictivity analysis, which requires the consideration of the prevalence of the studied population, we used the AS as a further comparison group, because this was a group with low seroprevalence. This is because these participants were less exposed to COVID-19 infection than HCWs and many of them had been in work-from-home arrangements for two days a week from 9 March 2020.

As mentioned above, participants that will test positive for SARS-CoV-2 specific antibodies, with at least one of the serological tests used in the study, will sample for NOS testing within 48 h after positive serological test results will be available. RT-PCR testing on NOS samples will perform using the Seegene Allplex™ 2019-nCoV assay, and a positive result (i.e., a Ct less than 40) for at least one of two viral targets (i.e., RdRP and N genes) indicated the presence of SARS-CoV-2 RNA. As current studies show marked variation and are likely to overestimate sensitivity, we used the lower end of current estimates from systematic reviews, with the approximate numbers of 70% for sensitivity and 95% for specificity, for illustrative purposes.

Descriptive analysis will perform for sex, age, professional category, and wards of the HCWs. The difference between proportions will evaluate with the two proportion Z test. Seroprevalence will calculate, separately, for tests on the venous samples and the POC tests. Seroprevalence for the tests on the venous samples will estimate as the proportion of individuals who will have a positive result of IgG in the immunoassay. Furthermore, for the tests on capillary blood, seroprevalence for both IgM and IgG will estimete as the proportion of individuals who will have positive results in the corresponding band of the POC test.

We also re-estimate the sensitivity and specificity of the POC test using the immunoassay as a reference. The accuracy of the capillary versus the venous test will evaluate with sensitivity, specificity, and predictive values with 95% confidence intervals (CIs). Each of the seroprevalences will stratify for professional category, age, and wards in which they worked during the COVID-19 emergency.

The difference between positivity in one of the serological tests and positivity in the RT-PCR on NOS samples will estimate through Pearson's chi-squared tests. The Spearman rank test (Bonferroni-adjusted) will use to evaluate the correlation between the anti-SARS-CoV-2 IgG assay in capillary blood versus the same titer in venous blood.

ELIGIBILITY:
Inclusion Criteria:

* employees of the Fondazione Policlinico Gemelli Hospital

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: medical, non-medical HCW, and administrative staff (AS) of the Fondazione Policlinico Gemelli Hospital
Sampling Method: Non-Probability Sample
Enrollment: 4888 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Detection of Anti-SARS-CoV-2 Antibodies in Blood Samples | 1 month
  Prevalence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection based on the serological tests and stratified by age, sex, professional category, and direct assistance to COVID-19 patients or not (COVID-19 care, Yes/No)

SECONDARY OUTCOMES:
Number of Healthcare Workers with Confirmed COVID-19 Infection | 1 month
  This outcome measure will track the number of healthcare workers who have a confirmed diagnosis of COVID-19. Confirmation will be based on positive PCR tests for detecting SARS-CoV-2.
Sensitivity and Specificity of Serological Tests | 1 month
  This outcome measure will assess the performance of serological tests in detecting antibodies to SARS-CoV-2 by calculating the sensitivity (the percentage of true positives correctly identified) and specificity (the percentage of true negatives correctly identified).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No